CLINICAL TRIAL: NCT03085589
Title: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Amulet Technology Development & Validation
Brief Title: MOWI Amulet Mobile Health Technology Validation
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, John A. Batsis, MD, Associate Professor of Medicine and of The Dartmouth Institute Geisel School of Medicine at Dartmouth, Dartmouth-Hitchcock Medical Center
Other Study IDs: D16182_1b; K23AG051681 (NIH)
Record Dates: First submitted 2017-02-27; First posted 2017-03-21 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Obesity
Keywords: elderly; telemedicine; obesity; rural health; health promotion
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Amulet adaptation and validation: The Amulet development team will develop and configure applications assessing: steps/distance; strength; activity type; gait speed; and real-time, self-monitored activity feedback. Objective measures will be validated with the Amulet from 60 participants ensuring usability and feasibility. Each participant will be asked to come into the clinic for one afternoon for about 2-3 hours.

SUMMARY:
This study aims to adapt a mobile health device (Amulet) for use in older adults. It is the second in a series of four research studies whose overarching goal is to conduct a program of pilot research aimed at developing and evaluating a technology-assisted wellness intervention for older adults with obesity who may or may not live in a rural area.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-64; and Age≥65 years
* Body Mass Index (BMI) ≥ 30kg/m^2 for those aged≥65 years
* Waist circumference ≥88cm in females or ≥102cm in male for those aged≥65 years

Exclusion Criteria for those aged ≥65 years:

* Severe mental or life-threatening illness
* Dementia
* Substance use
* History of bariatric surgery
* Suicidal ideation
* Unable to perform measures
* Reside in nursing home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants screened and recruited primarily in local primary care setting (Department of Community and Family Medicine at Dartmouth Hitchcock Medical Center), as well as through other marketing channels such as posters and radio advertising. Community leaders and clinicians recruited by invitation from the principal investigator.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Step Count Reliability | All outcomes of this Aim will take approximately 3 hours
  Assessment of step counts using Amulet application and validate this based on observation.
Strength Reliability | All outcomes of this Aim will take approximately 3 hours
  Assessment of strength using Amulet-based Therabands and validated against a dynamometer
Sit-to-Stand Reliability | All outcomes of this Aim will take approximately 3 hours
  Assessment of sit-to-stand Amulet application validated against a conducted test
Activity Reliability | All outcomes of this Aim will take approximately 3 hours
  Assessment of activity application validated against observations

SECONDARY OUTCOMES:
Satisfaction of Amulet | All outcomes of this Aim will take approximately 3 hours
  Participants will be asked to respond to questions regarding usability of the Amulet mobile device measured using a Likert scale

CONTACTS AND LOCATIONS:
Overall Officials: John A Batsis, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center / Dartmouth Medical School
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Qualitative Assessment — https://clinicaltrials.gov/ct2/show/NCT03041831
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Research Pilot — https://clinicaltrials.gov/show/NCT03104192
- See also: Mobile Health Obesity Wellness Intervention in Rural Older Adults (MOWI): Home-Based Pilot — https://clinicaltrials.gov/show/NCT03104205

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/89/NCT03085589/Prot_SAP_ICF_000.pdf